CLINICAL TRIAL: NCT03703388
Title: A Phase I Single-arm Dose Escalation Study to Determine the Safety and Bioavailability of a Natural Compound Arctigenin in Healthy Men
Brief Title: The Safety and Intake Rate of a Natural Compound Arctigenin in Healthy Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Charles Drew University of Medicine and Science (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Professor of Medicine, University of California, Los Angeles
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: IRB#: 18-000639
Record Dates: First submitted 2018-10-09; First posted 2018-10-12 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Healthy
MeSH Terms: interventions — arctigenin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arctigenin 250mg (Experimental): Arctigenin 250mg will be administered for 28 days.
  Interventions: Dietary Supplement: Arctigenin
- Arctigenin 400mg (Experimental): Arctigenin 400mg will be administered for 28 days.
  Interventions: Dietary Supplement: Arctigenin
- Arctigenin 500mg (Experimental): Arctigenin 500mg will be administered for 28 days.
  Interventions: Dietary Supplement: Arctigenin

INTERVENTIONS:
Dietary Supplement: Arctigenin — Arctigenin capsule

SUMMARY:
The purpose of this research study is to determine if consuming arctigenin, a natural compound from a Chinese herb called Arctium lappa (commonly called greater burdock), is safe, and to measure the intake level of arctigenin in blood. Arctigenin is being studied by researchers for potential health benefits such as helping to lower the risk of inflammation and cancer. A human study has been done measuring the uptake of arctigenin into blood after consumption of the herb extract containing arctigenin, and found no toxicity. Studies in mice demonstrated that consumption of arctigenin in pure form at a safe level is highly effective in inhibition of prostate cancer growth. Therefore, this study is designed to evaluate the safety and uptake rate of pure arctigenin in humans, which may be potentially used in the future for prostate cancer prevention.

DETAILED DESCRIPTION:
Phytochemicals are bioactive natural compounds extracted from plants. Phytochemicals have been considered as a major resource for developing non-toxic agents in prevention and treatment of chronic diseases, such as diabetes and cancer. However, most phytochemicals have low absorption rates, and the dose levels necessary for their beneficial effects can barely be achieved in the body after oral consumption, which limits their effect in humans. Therefore it is in urgent need to identify phytochemicals of higher uptake rate (or termed bioavailability). Arctigenin is a novel anti-inflammatory lignan mainly existing in the seeds of the herb Arctium lappa. This herb particularly its seeds has been widely used in traditional Chinese medicine to treat inflammation-related diseases such as cold, sore throat, and cough. The anti-cancer activity of arctigenin has recently been identified in cultured cancer cells and in animal models of several cancers. In prostate cancer, we found that arctigenin is highly effective in inhibition of the growth of cultured prostate cancer cells, while without affecting normal cells. The strong anti-tumor activity of arctigenin was further confirmed in our animal studies with prostate cancer mouse models. By analysis of blood concentrations of arctigenin, we found that the effective dose of arctigenin as observed in cultured cancer cells was achievable in mouse blood after consumption of arctigenin at a safe level, which suggests that the bioavailability of arctigenin is adequately high for its anti-cancer effect in organisms. We therefore propose a phase I one-arm dose escalation study to confirm the safety and bioavailability of arctigenin in healthy men, and to determine the dosage for future phase II studies in prostate cancer prevention. The study will use the traditional 3+3 design, which is the most widely used phase I design in oncology. Three dose levels of arctigenin will be tested, and participants will receive two capsules of arctigenin per day for 28 days, each capsule containing 250 mg of arctigenin. Initially there will be three participants on each dose level. If there is no dose-limiting toxicity (DLT) observed in any participant, the dose will be escalated to the next level. If DLT is observed in one or two participants, three more participants will be added. If DLT is observed in one or two participants out of the six, the dose will be escalated to the next level. If DLT is observed in three or more participants of the six, the previous dose level will be considered as the maximally tolerated dose (MTD), and three more patients will be added to the MTD group for a more accurate evaluation of the safety. The estimated MTD is the highest dose level with observed toxicity rate less than 0.33. Blood samples will be collected at baseline, during week 2 and on the last day of the study. Urine samples will be collected once a week during the intervention. On the last day of the intervention (Day 28) we will perform a single dose challenge with arctigenin and collect blood at baseline and at 1h, 2h, and 3h after arctigenin consumption in the morning. Arctigenin and its glucuronide will be analyzed in blood and urine using high performance liquid chromatography (HPLC)

ELIGIBILITY:
Inclusion Criteria:

1. Subjects consent to participate in the trial;
2. The subject is 20-75 years of age;
3. The subject is in healthy condition;
4. The subject agrees to stop consuming or using arctigenin-containing products and supplement throughout the entire intervention period except for arctigenin capsules provided during study intervention.

Exclusion Criteria:

1. History of hepatitis or liver dysfunction;
2. History of kidney disease or dysfunction;
3. Ongoing alcohol abuse;
4. Significant medical or psychiatric conditions that would make the patient a poor protocol candidate;
5. Prior sensitivity or allergic reaction to arctigenin-containing products or supplements;
6. Allergies to multiple food items or nutritional supplements;
7. Taking antibiotics, anti-diabetic medicines, anti-cancer medicine, LHRH agonists, androgen receptor blocking agents, finasteride, or has undergone bilateral orchiectomy.

Ages: 20 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Born male
Enrollment: 21 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 28 days
  To determine the maximum tolerated dose (or recommended dose) for future phase II studies by assessing the dose-limiting toxicities related to arctigenin consumption

SECONDARY OUTCOMES:
Bioavailability | 28 days
  2. To determine the bioavailability of arctigenin by measuring the concentrations of arctigenin and its glucuronide conjugates in serum collected before (T=0) and one hour (T1), two hours (T=2), and three hours (T=3) after the intake of a morning dose of arctigenin on Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Henning, PhD, Principal Investigator — University of California, Los Angeles; Piwen Wang, PhD, Principal Investigator — Charles Drew University of Medicine and Science
Locations (1):
- UCLA Center for Human Nutrition, 900 Veteran Avenue, WH 14-187, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No